CLINICAL TRIAL: NCT05692739
Title: Ensayo Clínico Para Determinar La Eficacia Y Seguridad Del Colirio De Insulina En El Tratamiento Del Ojo Seco En Pacientes Con Ojo Seco
Brief Title: Clinical Trial to Determine the Effectiveness and Safety of Topical Insulin in Dry Eye
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Barbara Burgos Blasco (Other)
Responsible Party: Sponsor-Investigator, Barbara Burgos Blasco, Ophthalmologist, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/211-EC_M
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye; Insulin
MeSH Terms: conditions — Dry Eye Syndromes; Insulin Resistance | interventions — Insulin; Cyclosporins; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial for the treatment of dry eye disease with three arms: topical insulin, topical cyclosporin (gold standard) and artificial tears (placebo)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Insulin (Experimental): Topical insulin 1UI/ml 4 times a day
  Interventions: Drug: Insulin
- Cyclosporin (Active Comparator): Cyclosporin 0,05% every 12 hours
  Interventions: Drug: Cyclosporins
- Artificial tears (Placebo Comparator): Artificial tears 4 times a day
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Insulin — see arm description
  Arms: Insulin
Drug: Cyclosporins — see arm description
  Arms: Cyclosporin
Drug: Artificial tears — see arm description
  Arms: Artificial tears

SUMMARY:
This is a parallel randomized controlled trial for the treatment of dry eye disease. The main objective is to investigate the efficacy and safety of the use of insulin eye drops in the control of moderate-severe dry eye disease. Topical insulin drops will be compared to the current gold standard treatment, cyclosporin and placebo (artificial tears).

DETAILED DESCRIPTION:
Patients will be recruited in Madrid. Patients with dry eye disease and no topical treatment other than artificial tears will be identified through the Ophthalmology clinic. They will be directly referred to a physician who is participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Dry eye disease diagnosis
* Treatment with artificial tears or hyaluronic acid gels for at least 3 months
* Signed informed consent by the patient
* Staining equal to or greater than Oxford II

Exclusion Criteria:

* Under 18 years old
* Corneal staining under Oxford II
* Treatment for dry eye disease other than artificial tears or hyaluronic acid gels
* Severe dry eye disease that requires immediate treatment
* Eye surgery in the last 6 months
* Other concomitant corneal pathology, eyelid malpositions, nasolacrimal drainage abnormalities, blinking alterations
* Contact lenses
* Other treatment besides artificial tears or hyaluronic acid gels
* Visual acuity less than 0.1
* Allergy or intolerance to any of the components included in the study
* Modifications in systemic immunosuppressive treatment
* Pregnancy or lactation
* Women of childbearing age who do not use a highly effective contraceptive method
* History of alcohol or drug abuse
* Participation in another clinical trial in the last 30 days
* Systemic pathology (cardiopulmonary pathology, connective tissue disorders, neurological or psychiatric pathology) or baseline situation of the patient that does not allow the examination (such as mental or psychomotor retardation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change of corneal staining from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Corneal staining will be evaluated on the slit-lamp and on slit-lamp images (masked evaluator)

SECONDARY OUTCOMES:
Changes in dry eye symptoms from baseline to 6 months after treatment time | From baseline to 6 months after treatment
  Dry eye symptoms will be evaluated using OSDI
Changes in esthesiometry from baseline to 6 months after treatment time | From baseline to 6 months after treatment
  Esthesiometry will be evaluated using an esthesiometer
Changes in tear rupture time from baseline to 6 months after treatment time | From baseline to 6 months after treatment
  Tear rupture time will be evaluated using the Keratograph (Oculus)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burgos Blasco, MD, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz-Valle D, Burgos-Blasco B, Rego-Lorca D, Puebla-Garcia V, Perez-Garcia P, Benitez-Del-Castillo JM, Herrero-Vanrell R, Vicario-de-la-Torre M, Gegundez-Fernandez JA. Comparison of the efficacy of topical insulin with autologous serum eye drops in persistent epithelial defects of the cornea. Acta Ophthalmol. 2022 Jun;100(4):e912-e919. doi: 10.1111/aos.14997. Epub 2021 Aug 18. PMID 34407296
- [Background] Diaz-Valle D, Burgos-Blasco B, Gegundez-Fernandez JA, Garcia-Caride S, Puebla-Garcia V, Pena-Urbina P, Benitez-Del-Castillo JM. Topical insulin for refractory persistent corneal epithelial defects. Eur J Ophthalmol. 2021 Sep;31(5):2280-2286. doi: 10.1177/1120672120958307. Epub 2020 Sep 21. PMID 32951459